CLINICAL TRIAL: NCT01785290
Title: Prophylactic Haloperidol Use for Delirium in ICU Patients; a Randomized Placebo-controlled Double-blind Multicentre Trial
Brief Title: pRophylactic halopEriDol Use for Delirium in iCu patiEnts With a High Risk for Delirium
Acronym: REDUCE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Delirium_Haldol-prophy; 2012-004012-66 (EudraCT Number); 2012/424 (Other: Medical Ethical Committee of Arnhem-Nijmegen)
Record Dates: First submitted 2013-01-31; First posted 2013-02-07 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2015-12

CONDITIONS: Delirium
Keywords: Delirium; Survival; Side-effects; QoL
MeSH Terms: conditions — Delirium | interventions — Haloperidol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Haloperidol 1mg/q8h (Experimental): Prophylactic haloperidol of 1 mg/q8h i.v.
  Interventions: Drug: Haloperidol 1 mg/q8h
- Haloperidol 2mg/q8h (Experimental): Prophylactic haloperidol 2mg/q8h i.v.
  Interventions: Drug: Haloperidol 2 mg/q8h
- Sodium chloride 0.9% (Placebo Comparator): Placebo (Sodium chloride 0.9%) three times a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol 1 mg/q8h — Patients receive prophylactic haloperidol until discharge from the ICU or when delirium occurs. In the latter case study drug will be stopped and patients will be subsequently treated according to the delirium protocol with open-label haloperidol. To avoid unnecessary risk for side-effects the dose will be halved in patients:
  * aged ≥ 80 years
  * weight ≤ 50 kg
  * liver failure
  Patients with an adjusted dosage of study drug remain allocated to their original group.
  In case of occurrence of QTc-time prolongation the study drug will be stopped. After normalisation of QTc-time (<500msec.) the study drug will be restarted. If QTc-time becomes prolonged again, the study drug will be stopped definitively. The patient will remain allocated to the original study group.
  Other Names: Haldol
  Arms: Haloperidol 1mg/q8h
Drug: Haloperidol 2 mg/q8h — Patients receive prophylactic haloperidol until discharge from the ICU or when delirium occurs. In the latter case study drug will be stopped and patients will be subsequently treated according to the delirium protocol with open-label haloperidol. To avoid unnecessary risk for side-effects the dose will be halved in patients:
  * aged ≥ 80 years
  * weight ≤ 50 kg
  * liver failure
  Patients with an adjusted dosage of study drug remain allocated to their original group.
  In case of occurrence of QTc-time prolongation the study drug will be stopped. After normalisation of QTc-time (<500msec.) the study drug will be restarted. If QTc-time becomes prolonged again, the study drug will be stopped definitively. The patient will remain allocated to the original study group.
  Other Names: Haldol
  Arms: Haloperidol 2mg/q8h
Drug: Placebo — Sodium Chloride 0.9%
  Other Names: Sodium Chloride 0.9%
  Arms: Sodium chloride 0.9%

SUMMARY:
The aim of this study is to determine the effects of a low dosage of prophylactic haloperidol in patients with a high risk to develop delirium, defined by an expected ICU length of stay of >1 day. The investigators hypothesized that haloperidol prophylaxis in patients with a high risk for delirium reduces 28-day mortality, delirium and delirium related outcome.

Two different dosages of haloperidol are used in this study to compare with placebo. A dosage of 1mg, or 2mg or placebo three times a day in a double-blinded fashion resulting in a three-armed multicentre randomized double-blinded placebo-controlled trial. To relate the potential beneficial effects of haloperidol to the a priori risk to develop delirium, the PREDELIRIC-model (delirium prediction model for ICU patients) will be used. This will enable the investigators to determine the preventive efficacy of haloperidol in patient groups based on their risk to develop delirium.

DETAILED DESCRIPTION:
In this study high risk patients will be included. Based on historical data the investigators know that the median predicted delirium risk is 35% in patients with an expected stay on the ICU of over one day. This is considered a high risk to develop delirium.

To assess patients for delirium using the Confusion Assessment Method (CAM)-ICU is part of daily clinical practice in all participating centres. In this study, high risk patients will receive three times a day a study drug of which two groups receive a low dose of haloperidol (1mg or 2mg) and a third arm will receive placebo.

This drug is worldwide the first choice of drug to treat delirious patients. When delirium is diagnosed, patients are treated according to delirium protocol, using a higher dosage than in the prophylactic treatment period as described in the study protocol. It is recognized that early treatment of delirium has beneficial effects compared with delayed treatment, and there is also some evidence that delirium prevention in ICU patients has beneficial effects, but the design of these previous studies was not optimal.

Potential side-effects of haloperidol include, extrapyramidal symptoms, drowsiness, agitation, and ventricular arrhythmias. The latter are extremely rare (only case-reports are published) and related to a higher dosage of haloperidol. With the dosage that will be used in the present study no relevant side-effects are anticipated. Nevertheless, and given the preventive nature of this study, extra attention is being paid on recognition of possible side-effects of haloperidol in the protocol. Importantly, in three recent prophylactic haloperidol studies no relevant side-effects, and in particular no ventricular arrhythmias, were reported using a similar low dosage of haloperidol as described in the present protocol.

During the study several inter-rater reliability checks (delirium experts versus ICU nurses) concerning the CAM_ICU assessments will be performed. Also medical and nursing files will be checked to secure the quality of the delirium diagnose.

The study will be monitored (all sites), randomly included patient data will be checked on delirium diagnose and endpoints of the study. All data will be collected by Electronic CRF. A check of completeness on all data is build-in.

All variables are defined using a data dictionary (using the NICE data dictionary) supplemented with definitions of PREDELIRIC-model predictors, delirium diagnosis (at least one positive CAM-ICU assessment), and delirium duration.

Sample size calculation is based on the effect on number of days of survival in 28-days mortality derived from the evaluation study using low dosage of prophylactic haloperidol. If the true hazard ratio of control patients relative to intervention patients is 0.85, taken into account an accrual time of 90 days with 28 days of follow-up, the investigators will need to study 647 patients per intervention group and 647 control patients to be able to reject the null hypothesis that the experimental and control survival curves are equal with probability (power) 0.80. The Type I error probability associated with this test of this null hypothesis is 0.05. Taken into account a drop out of 10% the investigators will include 715 patients per group; in total 2145 patients. The investigators assume that the effect on number of days of survival in 28-days mortality will be comparable between the two intervention groups. The Cox-regression analysis group will have three levels (placebo, 1 mg and 2 mg haloperidol three times daily).

A Data Safety Monitoring Board (DSMB)will monitor the safety of the study including interim analyses on safety/futility after 175-350 and 500 patients and safety and superiority after 1000 patients. Followed by a final analysis after 2145 patients.

Only for the interim analysis after 500 and 1000 patients adjusting for covariates (age, gender, delirium prediction score and sepsis) will be performed to determine the effect on 28-day survival

This multicenter study will be performed in:

* Radboud University Nijmegen Medical Centre
* University Medical Centre Utrecht
* Medical Centre Leeuwarden (stopped January 2014)
* Onze Lieve Vrouwen Gasthuis, Amsterdam (stopped March 2015)
* Isala Clinic, Zwolle (stopped June 2014)
* Canisius Wilhelmina Ziekenhuis, Nijmegen
* Medisch Spectrum Twente, Enschede
* Gelre Hospital, Apeldoorn
* Atrium Medical Centre, Heerlen
* Jeroen Bosch Hospital, Den-Bosch
* Atrium Medical Centre, Heerlen
* Medical Centre Haaglanden (Westeinde and Antoniushove), Den-Haag
* Bronovo Hospital, Den-Haag
* St. Jansdal Hospital, Harderwijk
* Maxima Medical Centre, Veldhoven
* University Medical Centre, Groningen
* Amphia Hospital, Breda
* VieCuri Hospital, Venlo
* Scheper Hospital, Emmen (stopped August 2016)
* Diakonessenhuis Hospital, Utrecht
* Haga Hospital, Den-Haag

After the 4th interim analysis the DSMB advised to drop on study arm due to effectivity and efficiency reasons. Since July 2015 the study has been continued with two study arms and the included numbers of patients is adjusted to 1800 patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* expected length of ICU stay of over one day

Exclusion Criteria:

* history of epilepsy, Parkinson's disease, hypokinetic rigid syndrome, dementia or alcohol withdrawal syndrome
* patients admitted to the ICU for neurological reasons (including post-resuscitation patients)
* patients treated with other anti-psychotics
* prolonged QTc-time (>500msec) or history of serious ventricular arrhythmia (in last 12 months)
* pregnancy/breast feeding
* delirious before ICU admission
* serious auditory or visual disorders
* ICU-stay ≤1 day
* unable to understand Dutch
* severely mentally disabled
* serious receptive aphasia
* moribund and not expected to survive 2 days
* known allergy to haloperidol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 28-day
  Number of days of survival in 28-days after inclusion.

SECONDARY OUTCOMES:
Delirium incidence during ICU stay | up to 28 days
  The onset of delirium during ICU admission
Number of delirium free days | 28 days
  Number of delirium and coma-free days in 28 days
Delirium related outcome during ICU stay | up to 28 days
  Time to successful extubation, incidence of re-intubation, incidence of ICU readmission, and incidence of unplanned removal of tubes and catheters during period of 28-days after inclusion of study, use of physical restraints
Determining efficacy in different risk groups | up to 28 days
  Determine the preventive efficacy of haloperidol in different patient groups based on the a priori risk to develop delirium: In patients with a predicted risk up to 50%, 50-70%, 70-90%, above 90% the effect of haloperidol will be determined
Side effects of haloperidol prophylaxis during prophylactic treatment | up to 28 days
  Evaluating the incidence of known side effects of haloperidol during the prophylactic treatment period
All cause mortality | 90 day
  Number of days of survival in 90-days after inclusion, survival analysis stratifying for delirium incidence will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Mark van den Boogaard, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre, Dept of Intensive Care Medicine
Locations (1):
- Radboud University Medical Centre, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
on request available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: available on request
Access Criteria: on request

REFERENCES:
- [Derived] Duprey MS, van den Boogaard M, van der Hoeven JG, Pickkers P, Briesacher BA, Saczynski JS, Griffith JL, Devlin JW. Association between incident delirium and 28- and 90-day mortality in critically ill adults: a secondary analysis. Crit Care. 2020 Apr 20;24(1):161. doi: 10.1186/s13054-020-02879-6. PMID 32312288
- [Derived] Heesakkers H, Devlin JW, Slooter AJC, van den Boogaard M. Association between delirium prediction scores and days spent with delirium. J Crit Care. 2020 Aug;58:6-9. doi: 10.1016/j.jcrc.2020.03.008. Epub 2020 Mar 25. PMID 32247156
- [Derived] van den Boogaard M, Slooter AJC, Bruggemann RJM, Schoonhoven L, Beishuizen A, Vermeijden JW, Pretorius D, de Koning J, Simons KS, Dennesen PJW, Van der Voort PHJ, Houterman S, van der Hoeven JG, Pickkers P; REDUCE Study Investigators; van der Woude MCE, Besselink A, Hofstra LS, Spronk PE, van den Bergh W, Donker DW, Fuchs M, Karakus A, Koeman M, van Duijnhoven M, Hannink G. Effect of Haloperidol on Survival Among Critically Ill Adults With a High Risk of Delirium: The REDUCE Randomized Clinical Trial. JAMA. 2018 Feb 20;319(7):680-690. doi: 10.1001/jama.2018.0160. PMID 29466591
- [Derived] van den Boogaard M, Slooter AJ, Bruggemann RJ, Schoonhoven L, Kuiper MA, van der Voort PH, Hoogendoorn ME, Beishuizen A, Schouten JA, Spronk PE, Houterman S, van der Hoeven JG, Pickkers P. Prevention of ICU delirium and delirium-related outcome with haloperidol: a study protocol for a multicenter randomized controlled trial. Trials. 2013 Nov 21;14:400. doi: 10.1186/1745-6215-14-400. PMID 24261644